CLINICAL TRIAL: NCT05826964
Title: Levels of Circulating Tumor DNA as a Predictive Marker for Early Switch in Treatment for Patients With Metastatic (Stage IV) Breast Cancer: A Phase 2 Randomized, Open-Label Study
Brief Title: Levels of Circulating Tumor DNA as a Predictive Marker for Early Switch in Treatment for Patients With Metastatic (Stage IV) Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Frances Valdes-Albini, Assistant Professor of Clinical Medicine, University of Miami
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20221297
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; ER-positive Breast Cancer; HER2-negative Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Cyclin-Dependent Kinase 4; Anastrozole; Letrozole; exemestane; palbociclib; ribociclib; abemaciclib; Fulvestrant; Sirolimus; TOR Serine-Threonine Kinases; Everolimus; Selective Estrogen Receptor Modulators; Tamoxifen; Phosphatidylinositol 3-Kinases; Alpelisib; Drug Therapy; taxane; eribulin; Capecitabine; Vinorelbine; elacestrant; Poly Adenosine Diphosphate Ribose; olaparib; talazoparib; capivasertib; Proto-Oncogene Proteins c-akt

STUDY DESIGN:
Intervention Model Description: The study will have the following 3 steps:
  1. Step 1: All patients (N=450 to 500) will be receiving standard of care (SOC) frontline treatment regimens.
  2. Step 2: A subset of patients in Step 1 (N=160) will be randomized to continue same treatment (Arm 1) or switch to new treatment (Arm 2).
  3. Step 3: A subset of patients in Arms 1 and 2 will be switched to new treatment at time of first clinical progression, which is either second-line treatment for patients in Arm 1 or third-line treatment for patients in Arm 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Step 2 Arm 1: No Modification of Therapy (Experimental): Participants in Step 2 Arm 1 will first undergo ctDNA monitoring in Step 1, providing blood samples for ctDNA testing at the following timepoints until a rise in ctDNA leading to a ratio (ctDNA result at time of assessment/ctDNA level at baseline) greater than (>) 1 occurs:
  * Cycle 1 day 1 (C1D1),
  * Day 30 (D30) post-treatment initiation (±3 days),
  * Day 60 (D60) post-treatment initiation (±3 days), and then
  * every 8-9 weeks (±1 week).
  Participants will have no change in standard of care therapy administered in Step 1.
  Interventions: Drug: AI+CDK4/6i; Drug: SERD+CDK4/6i
- Step 2 Arm 2: Early Switch in Therapy (Experimental): Participants in Step 2 Arm 2 undergo an early switch in standard of care therapy received in Step 1:
  * From AI+CDK4/6i in Step 1 to one of the following alternate endocrine therapies (ET) or chemotherapy:
    * SERD+CDK4/6i
    * mTOR Inhibitor + AI
    * mTOR Inhibitor+SERD
    * mTOR inhibitor + Selective estrogen receptor modulator
    * PI3K inhibitor + SERD
    * AKT inhibitor + SERD
    * Oral SERD
    * PARPi
    * Clinical Trial
    * Chemotherapy
  * From SERD+CDK4/6i in Step 1 to one of the following alternate ET or chemotherapy:
    * mTOR Inhibitor + AI
    * mTOR Inhibitor+SERD
    * mTOR inhibitor + Selective estrogen receptor modulator
    * PI3K inhibitor + AI
    * PI3K inhibitor + SERD
    * Oral SERD
    * PARPi
    * Clinical Trial
    * Chemotherapy
  Participants will receive this therapy for approximately 14 months.
  Interventions: Drug: AI+CDK4/6i; Drug: SERD+CDK4/6i; Drug: mTOR inhibitor + AI; Drug: mTOR inhibitor + SERD; Drug: mTOR inhibitor + Selective estrogen receptor modulator; Drug: PI3K inhibitor + SERD; Drug: PI3K inhibitor + AI; Drug: Chemotherapy; Drug: Oral SERD; Drug: PARPi; Drug: AKT inhibitor
- Step 3: Treatment for Patients in Arm 1 (Experimental): For participants who were randomized to Step 2 Arm 1 and experience first clinical progression. Participants will receive second-line treatment, having the option to change from their AI+CDK4/6i to SERD+CDK4/6i, or from SERD+CDK4/6i treatment to alternative endocrine therapy or chemotherapy. Therapy options for Step 3 are the same as listed for participants randomized to Step 2 Arm 2 and is administered standard of care.
  Participants will receive this therapy for approximately 6 months.
  Interventions: Drug: AI+CDK4/6i; Drug: SERD+CDK4/6i; Drug: mTOR inhibitor + AI; Drug: mTOR inhibitor + SERD; Drug: mTOR inhibitor + Selective estrogen receptor modulator; Drug: PI3K inhibitor + SERD; Drug: PI3K inhibitor + AI; Drug: Chemotherapy; Drug: Oral SERD; Drug: PARPi; Drug: AKT inhibitor
- Step 3: Treatment for Patients in Arm 2 (Experimental): For participants who were randomized to Step 2 Arm 2 and experience first clinical progression.
  Total participation duration is approximately 6 months.
  Interventions: Other: Step 3 Arm 2

INTERVENTIONS:
Drug: AI+CDK4/6i — Participants will receive standard of care one of three available AI therapies in combination with one of three available CDK4/6i therapies:
  * AI: Anastrozole, Letrozole or Exemestane
  * CDK4/6i: Palbociclib, Ribociclib or Abemaciclib
  Other Names: Aromatase Inhibitor (AI) + Cyclin dependent kinase 4 and 6 inhibitor (CDK4/6i); Anastrozole; Letrozole; Exemestane; Palbociclib; Ribociclib; Abemaciclib
  Arms: Step 2 Arm 1: No Modification of Therapy; Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: SERD+CDK4/6i — Participants will receive standard of care SERD therapy in the form of Fulvestrant, in combination with one of three one of three available CDK4/6i therapies:
  * SERD: Fulvestrant
  * CDK4/6i: Palbociclib, Ribociclib or Abemaciclib
  Other Names: Selective Estrogen Receptor Degrader (SERD) + CDK4/6i; Fulvestrant; Palbociclib; Ribociclib; Abemaciclib
  Arms: Step 2 Arm 1: No Modification of Therapy; Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: mTOR inhibitor + AI — Participants will receive standard of care mTOR inhibitor therapy (Everolimus) in combination with AI therapy (Exemestane) in Step 2 Arm 2 and Step 3. mTOR inhibitor + AI therapy administered as one of the available options for early switch from AI+CDK4/6i or SERD+CDk4/6i therapy in administered in Step 1.
  Other Names: Mammalian target of rapamycin (mTOR) inhibitor + Aromatase Inhibitor (AI); Everolimus; Exemestane
  Arms: Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: mTOR inhibitor + SERD — Participants will receive standard of care mTOR inhibitor therapy (Everolimus) in combination with SERD therapy (Fulvestrant), in Step 2 Arm 2 and Step 3. mTOR inhibitor + SERD therapy administered as one of the available options for early switch from AI+CDK4/6i or SERD+CDk4/6i therapy in administered in Step 1.
  Other Names: Everolimus; Fulvestrant
  Arms: Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: mTOR inhibitor + Selective estrogen receptor modulator — Participants will receive standard of care mTOR inhibitor therapy (Everolimus) in combination with selective estrogen receptor modulator therapy (Tamoxifen) in Step 2 Arm 2 and Step 3. mTOR inhibitor + Selective estrogen receptor modulator therapy administered as one of the available options for early switch from AI+CDK4/6i or SERD+CDk4/6i therapy in administered in Step 1.
  Other Names: Everolimus; Tamoxifen
  Arms: Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: PI3K inhibitor + SERD — Participants will receive standard of care one PI3K inhibitor therapy (Alpelisib), in combination with SERD therapy (Fulvestrant) in Step 2 Arm 2 and Step 3. PI3K inhibitor + SERD therapy administered as one of the available options for early switch from AI+CDK4/6i or SERD+CDk4/6i therapy in administered in Step 1.
  Other Names: Phosphoinositide 3-kinase (PI3K) inhibitor + SERD; Alpelisib; Fulvestrant
  Arms: Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: PI3K inhibitor + AI — Participants will receive standard of care a PI3K inhibitor therapy (Alpelisib), in combination with an AI therapy (Letrozole) in Step 2 Arm 2 and Step 3. PI3K inhibitor + AI therapy administered as one of the available options for early switch from SERD+CDk4/6i therapy in administered in Step 1.
  Other Names: Alpelisib; Letrozole
  Arms: Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: Chemotherapy — Chemotherapy administered standard of care as an alternative therapy in Step 2 Arm 2 and Step 3.
  Other Names: Taxane; Eribulin; Capecitabine; Vinorelbine
  Arms: Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: Oral SERD — Participants will receive standard of care oral SERD therapy (Elacestrant) in Step 2 Arm 2 and Step 3. Oral SERD therapy administered as one of the available options for early switch from AI+CDK4/6i or SERD+CDk4/6i therapy in administered in Step 1.
  Other Names: Elacestrant
  Arms: Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: PARPi — For participants with germline breast cancer gene (BRCA) mutation(s). Participants will receive standard of care PARPi (Olaparib or Talazoparib) therapy in Step 2 and Step 3.
  Other Names: Poly(ADP-ribose) inhibitor (PARPi); Olaparib; Talazoparib
  Arms: Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Drug: AKT inhibitor — For participants with tumors with one or more phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) or AKT serine/threonine kinase 1 (AKT1) or phosphatase and tensin homolog (PTEN) alterations. Participants in Step 2 and Step 3 will receive standard of care AKT inhibitor as an alternative therapy.
  Other Names: Capivasertib; Protein kinase B (AKT) Inhibitor
  Arms: Step 2 Arm 2: Early Switch in Therapy; Step 3: Treatment for Patients in Arm 1
Other: Step 3 Arm 2 — Participants will receive third-line treatment standard of care as per their treating physician's choice according to National Comprehensive Cancer Network (NCCN) guidelines.
  Arms: Step 3: Treatment for Patients in Arm 2

SUMMARY:
The majority of patients (pts) with breast cancer have hormone receptor positive (HR+) disease, and this holds true for pts with advanced breast cancer (ABC). Currently frontline therapy for pts with HR+ ABC is antihormonal therapy with an aromatase inhibitor or selective estrogen receptor degrader plus a CDK4/6i. The proposed trial is a randomized study to further evaluate the potential benefit of switching a frontline regimen at the time that a molecular signal, ctDNA, suggests progression prior to detection of clinical progression using standard methods. The purpose of this study is to determine whether switching treatment earlier in the disease process, based on molecular progression, will increase the amount of time that a patient's metastatic breast cancer is controlled compared to patients with metastatic breast cancer who receive treatment later based on diagnostic imaging results or other methods currently used in medical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women age ≥ 18 years.
2. Patients with a diagnosis of ER+, human epidermal growth factor receptor 2 negative (HER2-) metastatic (Stage IV) breast cancer. Positivity status is defined as >10% staining for ER and immunohistochemistry (IHC) 0+ or IHC 1 or 2+ staining for HER-2, and fluorescence in situ hybridization (FISH) negative with standard pathology staining methods.
3. Patients with de novo metastatic disease at the Screening Visit must undergo a SOC diagnostic biopsy.
4. Archived tumor tissue available.
5. Women and men with proven locally advanced, locoregionally recurrent or metastatic disease adenocarcinoma of the breast not amenable to curative therapy. Note: patients relapsing while on adjuvant tamoxifen or AI are eligible for this study.
6. No prior systemic anticancer therapy for metastatic or advanced disease (chemotherapy targeted therapy or endocrine therapy (ET)).

   Note 1: prior endocrine therapy in the metastatic setting is not allowed unless initiated <30 days from study initiation or Cycle 1, Day 1 (C1D1).

   Note 2: prior initiation of luteinizing hormone-releasing hormone (LHRH) agonist or bone-directed agents, however, is allowed.
7. No visceral crisis. Visceral crisis is defined as advanced, symptomatic, visceral spread that is at risk of life-threatening complication in the short term and that requires chemotherapy.
8. Adequate organ and marrow function as defined below:

   * Hematological

     * Absolute neutrophil count (ANC) ≥1,500 cells/mm³
     * Platelets ≥100,000 cells/mm³
     * Hemoglobin ≥9.0 g/dL or ≥8.0 g/dL for patients with bone metastases and/or menstruating females with evidence of iron deficiency
   * Renal

     * Serum creatinine or Measured or calculated creatinine clearance (glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl)) ≤ 1.5 x upper limit of normal (ULN) or CrCl ≥ 40 mL/min. CrCl should be calculated per institutional standard.
   * Hepatic

     * Serum total bilirubin < 1.0 ULN
     * Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine transaminase (ALT) (serum glutamic-pyruvic transaminase (SGPT)). Aminotransferase (AST and ALT) ≤ 2.5 x ULN or 5 X ULN for patients with liver metastases
     * Albumin ≥ 2.5 mg/dL
9. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST V.1.1) or non-measurable disease that is evaluable.
10. Patients with an Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
11. Ability to understand and the willingness to sign a written informed consent document.
12. Life expectancy >3 months.
13. Postmenopausal women, women with suppressed ovarian function, or premenopausal women, provided they are being treated with monthly LHRH analogues and are willing to continue to receive LHRH agonist therapy for the duration of the trial. Menopausal patients or patients with suppressed ovarian function are defined as follows:

    * Women with bilateral oophorectomy
    * Postmenopausal women, as defined by any of the following criteria:

      * Age 60 or over
      * Age 50-59 years and meets the following criterion:
      * Amenorrhea for ≥12 months and follicle-stimulating hormone and estradiol levels within the postmenopausal range
      * Women with hysterectomy or chemotherapy-induced amenorrhea. Note: Patients with hysterectomy or chemotherapy-induced amenorrhea must display follicle stimulating hormone and estradiol levels within the postmenopausal range.
14. Resolution of all acute toxic effects from prior anticancer therapy or surgical procedures as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V 5.0 to grade 1 (except alopecia or other toxicities not considered a safety risk for the patient at Investigator's discretion)

Exclusion Criteria:

1. Patients who are currently receiving or have received treatment for a secondary cancer other than resected non-melanoma skin cancer lesions or in situ cancer within the past 24 months.
2. Prior exposure to CDK4/6i ≤12 months prior to enrollment.
3. Use of investigational drugs ≤28 days prior to study enrollment and during the study.
4. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or that makes participation in the trial to be not in the best interest of the patient in the opinion of the Investigator.
5. Locally advanced breast cancer or locoregional relapse amenable for any treatment with curative intent.
6. HER2+ or equivocal tumor status either on the primary or on the recurrent tumor defined as IHC 3+, FISH/chromogenic in situ hybridization (CISH) amplified or FISH/CISH equivocal according to the American Society of Clinical Oncologists (ASCO) 2015 criteria.
7. Prior endocrine therapy in the metastatic setting is not allowed unless initiated < 30 days from study initiation or Cycle 1, Day 1 (C1D1).
8. Prior treatment with any CDK 4/6 inhibitor in the metastatic setting is not allowed.
9. Any major surgery (defined as requiring general anesthesia) or significant traumatic injury within 4 weeks of treatment; however, surgical diagnostic procedure is allowed (even if under general anesthesia).
10. Known active, bleeding diathesis.
11. Any serious known concomitant systemic disorder incompatible with the study (at the discretion of the Investigator).
12. Patients unable to swallow tablets.
13. History of malabsorption syndrome or other condition that would interfere with enteral absorption.
14. Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated with local therapy (e.g., radiotherapy, stereotactic surgery) and are clinically stable and off anticonvulsants and steroids for at least 4 weeks before treatment initiation.
15. Known hypersensitivity to letrozole, anastrozole, exemestane, fulvestrant, or CDK4/6i or any of their excipients.
16. Uncontrolled electrolyte disorders that can compound the effects of a corrected QT (QTc) interval prolonging drug (eg, hypocalcemia, hypokalemia, hypomagnesaemia).
17. Patients treated within the last 7 days prior to treatment start in the study with medications that are known to be cytochrome (CYP) CYP3A4 inhibitors or drugs that are known to be CYP3A4 inducers.
18. Patients requiring palliative radiation within the 30 days following C1D1 in Step 1.
19. Patients already included in another therapeutic trial evaluating an investigational medicinal product or having received an investigational medicinal product within 3 months.
20. Any stage II, III, or IV cancer within 5 years preceding patient enrollment in the trial; however, multiple breast cancers (contralateral/ipsilateral cancers/local relapses) are allowed pending all tumor masses were ER+.
21. Any history of hematologic malignancy.
22. Pregnancy or lactation period. Women of childbearing potential must implement adequate nonhormonal contraceptive measures (barrier methods, intrauterine contraceptive devices, sterilization; LHRH agonist cannot be considered as an efficient contraceptive measure) during study treatment and for 90 days after discontinuation. A serum pregnancy test must be negative in premenopausal women or women with amenorrhea of less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival 1 (PFS1) Among Participants in Step 2 | Up to 36 months
  PFS1 is defined as the elapsed time in months from the date of randomization (at time a rise in ctDNA ratio > 1 is detected prior to clinical progression) to the date of first clinical progression or death as determined by standard clinical methods or death in randomized participants.

SECONDARY OUTCOMES:
Number of participants in Step 1 with rising ctDNA ratio > 1 | Up to 36 months
  The number of participants with rising circulating tumor DNA (ctDNA) ratio > 1 and no synchronous clinical progression in Step 1 will be reported.
Percentage of participants in Step 1 with rising ctDNA ratio > 1 | Up to 36 months
  The percentage of participants with rising ctDNA ratio > 1 and no synchronous clinical progression in Step 1 will be reported.
Time from enrollment to rise in ctDNA ratio > 1 for Participants in Step 1 | Up to 36 months
  The time measured in months from enrollment to rise in ctDNA ratio > 1 in participants in Step1 without synchronous clinical progression will be reported.
Overall Response Rate (ORR) Among Participants in Step 2 | Up to 36 months
  The overall response rate (ORR) will be defined as the percentage of participants achieving best response of complete response (CR) or partial response (PR) to protocol therapy. Response will be assessed by treating physician using the revised Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
Clinical Benefit Rate (CBR) Among Participants in Step 2 | Up to 36 months
  The clinical benefit rate (CBR) is defined as the percentage of patients with best treatment response of complete response (CR), partial response (PR), or stable disease (SD) will be reported. Response will be assessed by treating physician using the revised Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
Progression-Free Survival 2 (PFS2) Among Participants in Step 3 | Up to 36 months
  PFS in Step 3, which will be called PFS2, and is defined as the elapsed time in months from the date of randomization in Step 2 to date of second clinical progression or death during Step 3.
Progression-Free Survival 3 (PFS3) Among Participants in Step 3 | Up to 36 months
  PFS in Step 3, which will be called PFS2, and is defined as the elapsed time in months from the date of first clinical progression in Step 2 to date of second clinical progression or death during Step 3.
Overall Response Rate (ORR) Among Participants in Step 3 | Up to 36 months
  The overall response rate (ORR) will be defined as the percentage of participants in Step 3 achieving best response of complete response (CR) or partial response (PR) to protocol therapy. Response will be assessed by treating physician using the revised Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
Clinical Benefit Rate (CBR) Among Participants in Step 3 | Up to 36 months
  The clinical benefit rate (CBR) is defined as the percentage of patients in Step 3 with best treatment response of complete response (CR), partial response (PR), or stable disease (SD) will be reported. Response will be assessed by treating physician using the revised Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Valdes-Albini, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No